CLINICAL TRIAL: NCT03353714
Title: The Effect of Pudendal Blocks on Voiding Dysfunction Following Slings
Acronym: PUBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Flynn (Other)
Responsible Party: Sponsor-Investigator, Michael Flynn, MD, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H00013722
Record Dates: First submitted 2017-11-04; First posted 2017-11-27 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pudendal block with saline (Placebo Comparator): Pudendal block with normal saline
  Interventions: Other: Pudendal block
- Pudendal block with bupivacaine (Active Comparator): Pudendal block with bupivacaine
  Interventions: Other: Pudendal block

INTERVENTIONS:
Other: Pudendal block — Pudendal block with normal saline (for control group) and bupivacaine (for intervention group)

SUMMARY:
To determine the effect of a bilateral pudendal block on voiding dysfunction following midurethral slings.

DETAILED DESCRIPTION:
Midurethral slings (MUS) are commonly performed to treat stress urinary incontinence in women. One common complication is short-term postoperative voiding dysfunction. Approximately 20% of patients undergoing MUS have difficulty voiding in the immediate postoperative period and are discharged home with an indwelling bladder catheter. A pudendal block provides analgesia to the vulva, vagina, and perineum and is used in various fields, ranging from obstetrical indications to hemorrhoidectomies. The colorectal literature has demonstrated an improvement in postoperative voiding dysfunction with intraoperative bilateral pudendal blockade, presumably due to pain relief. However, only one study has explored the effect of a pudendal blockade on postoperative voiding in patients undergoing MUS. This was a small French case series of 9 patients, and it concluded that it was a safe procedure with good patient satisfaction. Given the scant literature evaluating voiding dysfunction following pudendal blocks in MUS, and the encouraging data from anorectal surgeries, we aim to study this effect via a randomized, placebo-controlled, double-blinded trial.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing a midurethral sling without concomitant procedures under general anesthesia

Exclusion Criteria:

* Unable to consent (lacking capacity)
* Under 18 years of age
* Pregnant women
* Prisoners
* Using intermittent self-catheterization preoperatively
* Neurological disease or spinal cord injury resulting in voiding dysfunction
* Allergy to bupivacaine
* Diagnosis of chronic pain syndromes
* Daily use of narcotics
* Intra-operative bladder injury necessitating use of a prolonged indwelling Foley catheter

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Postoperative voiding dysfunction | Prior to discharge home (within 24 hours)
  Postoperative void trial (discharge home with or without Foley catheter)

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Maheshwari, DO, Principal Investigator — UMass Medical School; Michael K Flynn, MD, Principal Investigator — UMass Medical School
Locations (1):
- University of Massachusetts, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article after de-identification.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Derived] Maheshwari D, Sierra T, Leung K, Hall C, Flynn M. Effect of Pudendal Blockade on Bladder Emptying After Midurethral Sling: A Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):e465-e468. doi: 10.1097/SPV.0000000000000963. PMID 33009265